CLINICAL TRIAL: NCT06717464
Title: Toripalimab Combined With Capecitabine as Postoperative Adjuvant Therapy for Patients With Resectable Advanced Extrahepatic Biliary Tract Cancer, Phase II, Single-center, Randomized Controlled Trial
Brief Title: Toripalimab Combined With Capecitabine as Postoperative Adjuvant Therapy for Patients With Resectable Advanced Extrahepatic Biliary Tract Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E20241189
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-10

CONDITIONS: Gallbladder Cancer; Hilar Cholangiocarcinoma; Distal Cholangiocarcinoma
MeSH Terms: conditions — Gallbladder Neoplasms; Klatskin Tumor | interventions — Capecitabine; toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Capecitabine therapy group (Experimental)
  Interventions: Drug: Capecitabine
- Toripalimab combined with capecitabine therapy group (Experimental)
  Interventions: Drug: Capecitabine; Drug: Toripalimab

INTERVENTIONS:
Drug: Capecitabine — 1250mg/m2, D1-D14, q3w, for 24 weeks (8 cycles)
Drug: Toripalimab — 240mg intravenous injection, q3w, for 54 weeks (18 cycles)
  Arms: Toripalimab combined with capecitabine therapy group

SUMMARY:
This is a randomized controlled study to evaluate the efficacy and safety of toripalimab plus capecitabine as postoperative adjuvant therapy for patients with resectable advanced extrahepatic biliary tract cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Both men and women aged ≥18 years old were eligible.
2. After radical surgery, postoperative pathological diagnosis of gallbladder cancer and Distal cholangiocarcinoma. TNM staging Ⅱ and above.
3. No systemic treatment before to participate in research;
4. ECOG PS score 0-1 points;
5. The main viscera function is normal, no serious blood, heart, lung, liver, kidney and bone marrow dysfunction, and immune deficiency disease.
6. Laboratory tests meet the following requirements: women of childbearing age must be within 14 days before the group for a pregnancy test results were negative serum or urine, and voluntary in the observation period and the last 8 weeks after with the study drug to adopt the appropriate methods of contraception; In men, either surgical sterilization or consent to use an appropriate method of contraception during the observation period and for 8 weeks after the last dose of the study drug was given.
7. Patients volunteered for and sign the informed consent;
8. Expect good adherence, can according to the plan calls for follow-up curative effect and adverse reactions.

Exclusion Criteria:

1. Postoperative pathology showed Pancreatic cancer and ampullary cancer;
2. The former group received PD 1, PD - L1, PD patients treated L2, CTLA 4, or directly to another stimulus or common weak T cell receptors (such as CTLA - 4, 0 x40, CD137) patients;
3. Use of any other study medication within 4 weeks before enrollment;
4. Have any active autoimmune disease or a history of autoimmune disease (e.g., interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (eligible after hormone replacement therapy)); Patients with complete remission of childhood asthma without any intervention in adulthood or with white scarring were eligible, but those requiring medical intervention with bronchodilators were not eligible;
5. People with innate or acquired immune deficiency, such as people with human immunodeficiency virus (HIV) infection;
6. Patients with uncontrolled cardiac clinical symptoms or diseases, such as unstable angina pectoris with NYHA II or higher heart failure, myocardial infarction within 1 year, clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention;
7. Severe infection (e.g., requiring intravenous antibiotics, antifungal, or antiviral drugs) within 4 weeks before the first dose, or unexplained fever >38.5°C during screening/before the first dose;
8. Known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
9. Live attenuated vaccine is administered within 4 weeks before the first dose or is planned for the duration of the study;
10. Patients with or accompanied by other systemic malignant tumors within the last 5 years (except cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and ovarian cancer);
11. Known allergy to any of the trial drugs;
12. Pregnant, lactating women and subjects with reproductive capacity were unwilling to take effective contraceptive measures;
13. Suffering from uncontrollable psychosis; fourteen Other conditions that the investigator deemed inappropriate for inclusion. If the patient has central nervous system metastasis, serious laboratory abnormalities, accompanied by family or social factors, it will affect the safety of the subject, or the collection of data and samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2024-11-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival rate | 1 year

SECONDARY OUTCOMES:
1-year OS | 1 year
2-year OS | 2-year
Occurrence of adverse reactions | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No